CLINICAL TRIAL: NCT07205354
Title: Design of a Food Preference Assessment Tool for Older Patients in Geriatrics Units
Brief Title: Design of a Food Preference Assessment Tool for Older Patients in Geriatrics units_DYSPHAGING-PREFERENCES
Acronym: DYSPHAGING-PRE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0022
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hospitalisation in Geriatrics; Swallowing Disorder; Eating Habits
Keywords: geriatric; denutrition; Dysphagia
MeSH Terms: conditions — Deglutition Disorders; Feeding Behavior | interventions — Acclimatization; Reproducibility of Results; Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Step 1: adaptation of the CFTQP to a geriatric population: This step was designed to assess the recognition of pre-selected food pictures in the older population. A group of at least 35 patients who have completed the entire questionnaire is expected.
  Interventions: Other: ADAPTATION
- Step 2: test-retest reliability analysis of the device: This step was designed to ensure individual reproductibility of the device. A group of at least 35 patients who have completed the entire questionnaire is expected.
  Interventions: Other: test-retest reliability
- Step 3: cross-sectional study: A group of at least 209 patients (including 35 patients of step 2) is expected
  Interventions: Other: Cross-sectional study

INTERVENTIONS:
Other: ADAPTATION — For each patient (set of at least 35 patients), the assessor will ask the patient:
  * Have you ever eaten this food? YES or NO
  * Does the photo match the description? YES or NO
  * 20 photos of foods per category are provided (10 + 10)
  * If the foods tested are recognised (YES answer to both questions) by more than 80% of the study population, they will be retained.
  * The 16 foods (8+8) with the highest recognition rates will be retained.
  * If fewer than 16 foods (8+8) per category are recognised, the list will be modified by retaining the recognised foods and adding new foods to obtain the 'modified list'.
    2- If the criteria are not validated, a modified list is resubmitted to a new sample of 35 patients until the objectives are validated and a suitable questionnaire is obtained.
  Obtaining an ADAPTED DYSPHAGING PREFERENCES QUESTIONNAIRE is a prerequisite for moving on to the test-retest reliability phase
  Groups: Step 1: adaptation of the CFTQP to a geriatric population
Other: test-retest reliability — For each patient (new set of 35 patients)
  * the DYSPHAGING preferences questionnaire (including previously adapted pictures) will be assessed and preference indexes will be determined.
  * Within 3-7 days, each patient will be asked for the forced choice in the second step of phase 2. A new preference index will be determined using the first recognition and the second forced choices answers.
  * Test-retest reliability will be assessed by determination of an intra-class correlation coefficient between the two indexes obtained for each patient tested. (Good test-retest reliability will be considered with an intra-class correlation coefficient upper than 0,75 in each category and will be expected in at least 4 of the 6 tested categories to perform the cross-sectional study (phase 3)
  Groups: Step 2: test-retest reliability analysis of the device
Other: Cross-sectional study — For each patient (new set of 174 patients)
  * the DYSPHAGING preferences questionnaire (including previously adapted pictures) will be assessed and preference indexes will be determined.
  * In addition, for each patient, collection of geriatric covariates obtained in routine care will be performed for analyses ( demographic characteristics (age, sex, functionality according to the activity of daily living (ADL)8 and instrumental ADL6 scores), local and factors affecting taste, mastication or dietary patterns (dental condition/dental apparatus, alcoholism, smoking, food allergies, comorbidities, treatments), nutritional status (ideal and current weight/height/BMI, albumin, pre-albumin, Vitamins B12, B9, D), comedications (as described as according to the galenic form and drug class prescribed) and swallowing disorders (EAT-10 score with cut-off of 3)
  Groups: Step 3: cross-sectional study

SUMMARY:
Swallowing disorders - or oral dysphagia (OD) - are identified as a cause of malnutrition. They gradually lead patients to withdraw certain foods from their diet, leading to progressive dietary imbalances, or increased cardiovascular risks. Two European societies (the European Society for Swallowing Disorders and the European Union Geriatric Medicine Society) have defined recommendations that include raising awareness of OD, the use of screening scores, preventive measures, diagnostic standardization and interventions implemented (re-education, adaptation of textures). We recently reported the results of the DYSPHAGING Pilot Study that validated the feasibility of a standardized care path including a systematic screening of OD and the implementation of preventive measures in geriatric wards.

DYSPHAGING Preferences is a three-step research program designed to develop (step 1) a specific device to evaluate food preferences in geriatric populations, adapted from the CFTPQ, evaluate its test-retest reliability (step 2), and perform a cross-sectional study to explore individual differences within the older population depending on their geriatric characteristics and, among them, on the presence or not of OD (step 3).

DETAILED DESCRIPTION:
The World Health Organization (WHO) has made the healthy aging of the population a priority in the orientation of public policies for the period 2016-2030. Aging is associated with a progressive decline in various physiological functions that can lead to a gradual risk of sarcopenia, malnutrition, dysphagia, osteoporosis and frailty. Due to multiples etiologies and both morbidity and mortality consequences, the management of malnutrition is one of the main challenges in the older population.

Swallowing disorders - or oral dysphagia (OD) - are identified as a cause of malnutrition. They gradually lead patients to withdraw certain foods from their diet, leading to progressive dietary imbalances, or increased cardiovascular risks. Two European societies (the European Society for Swallowing Disorders and the European Union Geriatric Medicine Society) have defined recommendations that include raising awareness of OD, the use of screening scores, preventive measures, diagnostic standardization and interventions implemented (re-education, adaptation of textures). The investigators recently reported the results of the DYSPHAGING Pilot Study that validated the feasibility of a standardized care path including a systematic screening of OD and the implementation of preventive measures in geriatric wards.

Current recommendations for the treatment of undernutrition involve increasing energy and protein intake. Apart from the quantitative needs, qualitative properties of the food delivered are less emphasized. Some surveys in geriatric populations have shown increased preferences for fruits, vegetables and fish, and a reduction in the variety of dishes or the consumption of dairy and meat products. In subjects with swallowing disorders, preferences are mainly oriented towards adapted textures, like foods finely cut into small pieces. However, hedonic properties have rarely been evaluated, and the combination of dietary restriction with the consumption of texture-modified foods can lead older patients to nutritional deficiencies.

In this context, strategies are needed to better tailor food intakes to the preferences of geriatric patients. In adult populations, individual differences in texture and taste perceptions have been demonstrated and impacted food appreciation. In addition, and more specifically in an older population polypharmacy, smell, mood or cognitive disorders, OD are highly prevalent and may have an impact on such appreciation.

Some tools have been developed to evaluate food preferences in different specific populations, but most of them are IT-based and poorly adapted to vulnerable older patients, due to frequent praxis, cognitive or visual impairments. Another tool, the Child Food Texture Preference Questionnaire (CFTPQ), has been specifically developed for pediatric populations. The CFTPQ is based on forced-choice question methods, that are, sequential choices between alternative meal presentations previously identified by the participants. Such procedures are widely used in consumer preference assessment surveys and in geriatric populations to assess the food preferences of patients with poor appetites, representative of hospital populations In addition, several studies have shown a concordance between the choices made by patients and their actual food consumption. However, the meal presentations included in the CFTPQ are inappropriate for a geriatric population.

Based on CFPTQ developed by Laureati et al. 2020, the DYSPHAGING preferences questionnaire is using a forced-choice method. The device is divided into two-stages:

* A first stage of individual recognition in which the patient is asked to answer the following question "have you already eaten this product?" for each of the foods evaluated in each of the 6 categories.
* A second stage in which the same patient is asked to choose between two paired foods presented at the same time ("which one of the two presented products would you like to eat?").

Evaluation of preference will be defined using food preference index, as previously described by Laureati et al. 2020, and defined as follow:

PREFERENCE INDEX = [(Sum of scores of valid pairs/number of valid pairs) -1]x100

* Valid pair is considered when both foods have been previously recognized on the individual recognition part. A minimum of six valid pairs is requested for each category.
* Scores correspond to a numerical value: for each pair of foods compared, when the food in the category is prioritized by the participant, the pair is given a score of 2; otherwise, it is given a score of 1. For a food category, the scores for each pair are summed. Only valid pairs are considered for sum calculations.

DYSPHAGING Preferences is a three-step research program designed to develop (step 1) a specific device to evaluate food preferences in geriatric populations, adapted from the CFTPQ, evaluate its test-retest reliability (step 2), and perform a cross-sectional study to explore individual differences within the participant depending on their geriatric characteristics and, among them, on the presence or not of OD (step 3).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 70
* Patient hospitalised in the healthcare sector (CSG, SMR)
* Patient or patient under guardianship informed of the study and having expressed no objection to participating in the study
* Patient under guardianship whose guardian has been informed of the study and has expressed no objection to the patient's participation in the study.

Exclusion Criteria:

* Patient unable to complete the questionnaire.
* Patient unable to eat orally

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will include older patient identified either during their admission (in acute care and rehabilitation units) or during systematic assessments in long-term care units. Patients likely to participate in the study will be identified within the geriatric ward as part of their regular medical follow-up. Patients will be informed of the existence of the protocol by an investigating physician or a member of the local healthcare team. A non-opposition will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Adapting a tool for assessing food preferences in patients over 70 years of age hospitalised in geriatric wards, based on a paediatric tool for assessing food texture preferences. | 1 to 3 days
  Proportion of foods recognised among those offered (a food will be retained if the proportion is greater than 0.8). The tool will be considered suitable when each category contains 8 foods of interest and 8 opposing foods, i.e. 16 foods recognised by at least 80% of the patients tested.
Assessing the reproducibility of the food preference index | 7 to 10 days
  Evaluation of the reproducibility of the preference indices obtained between the two questionnaires (intraclass correlation coefficient).
Assessing the association between dysphagia and food preferences | 7 to 10 days
  The presence of dysphagia disorders will be defined by a score of ≥ 3 on the EAT-10 questionnaire.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Pierre GARRAUD Unité de Soins Médicaux et de Réadaptation, Lyon
  - Groupement hospitalier Sud Court Séjour de Gériatrie, Pierre-Bénite
  - Groupement hospitalier Sud Unité de Soins Médicaux et de Réadaptation, Pierre-Bénite